CLINICAL TRIAL: NCT06444906
Title: A Two-Part, Randomized Study of Dermacyte® Amniotic Wound Care Matrix for the Treatment of Diabetic Foot Ulcers (DFU)
Brief Title: A Two-Part, Randomized Study of Dermacyte® Amniotic Wound Care Matrix
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merakris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM-DFU-201
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Dermacyte Matrix (Active Comparator): Dermacyte Matrix will be applied topically in conjunction with SOC on a weekly frequency and dosed by square centimeters to match the ulcer surface area.
  Interventions: Device: Dermacyte Matrix
- Standard of Care (Other): SOC therapy will consist of weekly debridement of nonviable tissue as clinically indicated, saline-moistened non-occlusive dressing, weight off-loading to decrease pressure on extremity, aggressive treatment of infection and arterial revascularization if indicated.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: Dermacyte Matrix — The appropriate square centimeters of Dermacyte Matrix is applied directly to the target DFU that is free of debris and necrotic tissue. The Dermacyte Matrix will be applied at weekly intervals or for up to 10 applications.
  Arms: Dermacyte Matrix
Other: Standard of Care (SOC) — SOC therapy will consist of debridement of nonviable tissue, saline-moistened non-occlusive dressing, weight off-loading to decrease pressure on extremity, aggressive treatment of infection and arterial revascularization if indicated at weekly intervals or for up to 10 applications.
  Arms: Standard of Care

SUMMARY:
This is a multi-center, prospective, two-part, controlled study to determine the percentage of participants with complete ulcer closure of a target DFU at Week 12 following treatment with Dermacyte Matrix or SOC.

DETAILED DESCRIPTION:
This is a multi-center, prospective, two-part, controlled study to determine the percentage of participants with complete ulcer closure of a target DFU at Week 12 following treatment with Dermacyte Matrix or standard of care (SOC).

Part 1 of the study will enroll 20 participants to determine the percentage of participants with a complete ulcer closure following treatment with Dermacyte Matrix at Week 12.

In Part 2 of the study approximately 65 participants will be randomized 1:1 to receive Dermacyte Matrix or SOC for 12 weeks. The final sample size for Part 2 may be adjusted based on the effect size observed in Part 1 of the study.

For the purposes of this study, SOC therapy will consist of debridement of nonviable tissue, saline-moistened non-occlusive dressing, weight off-loading to decrease pressure on extremity, aggressive treatment of infection and arterial revascularization if indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Participant 18 years old or older
2. Type I or Type II diabetes mellitus
3. Participant has well controlled glucose levels, with HbA1c < 12% within 3 months of Dermacyte Matrix application
4. Participant has adequate lower extremity perfusion, with Ankle-Brachial Index > 0.8 (note: this is an ABI-equivalent, based on biphasic or triphasic color duplex - PVR or MRA. Diabetics often have peripheral vascular calcification or poorly compressible vessels resulting in abnormally high Ankle-Brachial Indices.) or dorsum transcutaneous oxygen test (TcPO2) > 30 mmHg. The presence of tibial and plantar pulses is preferred.
5. Willing and able to tolerate and maintain the required weight off-loading of the affected limb and perform necessary dressing changes
6. DFU is full thickness (Wagner Grade I or II)
7. Adults with a chronic non-healing DFU (at least 30 days but no longer than 52 weeks old) will be eligible for enrollment
8. Participant's ulcer size >0.5cm2 and < 20cm2 area post-debridement
9. Participant has plantar ulcers of greater than or equal to 4 weeks duration at presentation, unresponsive to standard wound care
10. Participant should have no evidence of unresolved gross soft-tissue infection or boney pathology (i.e. osteomyelitis)
11. Participant should have no evidence of underlying co-morbid conditions that would adversely affect wound healing such as: Cancer, Raynaud's syndrome, severe venous insufficiency or uncorrected arterial insufficiency, etc.
12. Participant should not be on medications that compromise healing: cytotoxic chemotherapeutics, etc

Exclusion Criteria:

1. Suspected or confirmed signs of infection of the study ulcer/limb including soft-tissue infection or osteomyelitis
2. Subjects who are currently receiving, or have received within 4 weeks prior to study entry agents known to impair or affect wound healing, including:

   1. Adriamycin (doxorubicin), bleomycin, sirolimus (Rapamune, rapamycin) and anti-TNF cytotoxic/immunosuppressive agents;
   2. Radiation therapy at the ulcer site;
   3. Other immunosuppressive agents.
3. Subjects presenting with:

   1. Charcot foot with a bony deformity
   2. Chopart's amputation
   3. Calcaneus ulcers
4. Subjects previously treated with amniotic membrane or any other advanced therapy at the target site for 1 month prior to enrollment
5. Subjects with evidence of skin cancer within or adjacent to the ulcer site.
6. History of bone cancer of the affected limb
7. Subjects who have significant arterial disease as determined by ABI, duplex Doppler sonography (PVR) or magnetic resonance angiography (MRA): Ankle-Brachial Index < 0.8 (note: this is an ABI-equivalent, based on biphasic or triphasic color duplex - PVR or MRA. Diabetics often have peripheral vascular calcification or poorly compressible vessels resulting in abnormally high ABIs); dorsum transcutaneous oxygen test (TcPO2) < 30 mmHg; absence of tibial or plantar pulses.
8. Subjects who have documented clinically significant medical conditions, which would impair wound healing. This includes:

   1. Renal impairment (creatinine >2.5 mg/dL);
   2. Hepatic impairment (2XULN);
   3. Hematological disorders (abnormities of formed elements);
   4. Neurologic disorders resulting in significant impairment of sensory and motor functions as judged by the investigator;
   5. Excessive lymphedema that could interfere with wound healing
   6. Subjects with signs and symptoms of cellulitis;
   7. Subjects with ulcers with sinus tracts associated with an ongoing infection;
   8. Subjects with active deep vein thrombosis;
   9. Subjects with uncontrolled diabetes, as demonstrated by increased HbA1C (> 12%);
   10. Immunocompromised subjects (e.g., lymphoma, AIDS, myelodysplastic disorders)
9. HBOT within 3 days of treatment visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of Dermacyte Matrix compared to SOC based on total wound closure | 12 weeks
  Wound healing will be assessed by observation of skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits at least 2 weeks apart.

SECONDARY OUTCOMES:
To determine the safety of Dermacyte Matrix compared to SOC | 12 weeks
  Safety will be assessed throughout the study. Adverse events will be recorded using the NCI Common Terminology Criteria for Adverse Events Version 5 (CTCAE v5).
To determine the heal rate of DFU for Dermacyte Matrix and SOC | 12 weeks
  Healing rate will be assessed by percent area reduction of the target ulcer from Baseline to Week 12.

OTHER OUTCOMES:
To measure change in quality of life (QoL) | 12 weeks
  QoL will be assessed at Baseline and Week 12 via patient reported outcomes using the Neuro-QoL (Quality of Life in Neurological Disorders); a disease-specific instrument that has been validated for assessing the impact of peripheral neuropathy and foot ulceration and quality of life in patients with diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Sean O'Connell, PhD, Study Director — Consultant

IPD SHARING:
Plan to Share IPD: No